CLINICAL TRIAL: NCT03610542
Title: Reducing Clinical Anxiety in Adolescents Through Selective Intervention
Brief Title: School-based Interventions for Test Anxiety in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Liverpool John Moores University (Other)
Collaborators: Wellcome Trust (Other); Manchester University (Unknown); Leeds University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHC0341
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Anxiety
Keywords: Test Anxiety; Wellbeing
MeSH Terms: conditions — Anxiety Disorders | interventions — Precipitating Factors; Organizational Objectives

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of three conditions: Cognitive behavioural therapy with no booster sessions, Cognitive behavioural therapy with 2 booster sessions or a no intervention control arm.
Who Masked: Participant
Masking Description: Sequentially numbered opaque sealed envelopes will be used to conceal allocation. Envelopes will be prepared by a member of the research team and opened by participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behaviour Therapy (Experimental): Cognitive behaviour therapy conducted in groups of 6-8 persons.One forty-five minute session per week for 6 weeks: Triggers for anxiety, identifying and challenging negative thoughts, relaxation, overcoming avoidance, and goal setting.
  Interventions: Behavioral: Triggers for anxiety; Behavioral: Identifying and challenging negative thoughts; Behavioral: Relaxation; Behavioral: Goal Setting; Behavioral: Overcoming avoidance
- Cognitive Behaviour Therapy with 2 Booster Sessions (Experimental): Cognitive behaviour therapy conducted in groups of 6-8 persons.One forty-five minute session per week for 6 weeks: Triggers for anxiety, identifying and challenging negative thoughts, relaxation, overcoming avoidance, and goal setting. 2 booster sessions (forty-five minutes each) will be provided at three and nine months. Each session will recap the content of the initial 6 sessions.
  Interventions: Behavioral: Triggers for anxiety; Behavioral: Identifying and challenging negative thoughts; Behavioral: Relaxation; Behavioral: Goal Setting; Behavioral: Overcoming avoidance
- Control (No Intervention): This is a no intervention control arm

INTERVENTIONS:
Behavioral: Triggers for anxiety — Students learn about different triggers for anxiety, what the signs and indicators of anxiety are, and identify their own triggers for anxiety
  Other Names: STEPS
  Arms: Cognitive Behaviour Therapy; Cognitive Behaviour Therapy with 2 Booster Sessions
Behavioral: Identifying and challenging negative thoughts — Students learn about the types of unrealistic thoughts that underpin anxiety and how anxiety can be reduced with more realistic thoughts. Students identify their own unrealistic thoughts that contribute to anxiety and what more realistic thoughts can be used.
  Other Names: STEPS
  Arms: Cognitive Behaviour Therapy; Cognitive Behaviour Therapy with 2 Booster Sessions
Behavioral: Relaxation — Students are taught to relax through (1) breathing exercises, (2) progressive muscle relaxation, and (3) imagery. Student practice these techniques.
  Other Names: STEPS
  Arms: Cognitive Behaviour Therapy; Cognitive Behaviour Therapy with 2 Booster Sessions
Behavioral: Goal Setting — Students learn how to set goals, monitor goal progress, and check when goals have been achieved. Students then identify their own goals.
  Other Names: STEPS
  Arms: Cognitive Behaviour Therapy; Cognitive Behaviour Therapy with 2 Booster Sessions
Behavioral: Overcoming avoidance — Students identify ways that they avoid anxiety-provoking situations (e.g., procrastinating exam study). Students develop plans for exposure to anxiety-provoking situations and learn study strategies to build confidence.
  Other Names: STEPS
  Arms: Cognitive Behaviour Therapy; Cognitive Behaviour Therapy with 2 Booster Sessions

SUMMARY:
This study evaluates the clinical and cost effectiveness of test anxiety as a form of selective prevention for clinical anxiety. Participants will be randomly allocated to cognitive behavioural therapy without booster sessions, cognitive behavioural therapy with two booster sessions, or a no intervention control.

DETAILED DESCRIPTION:
Test anxiety affects a substantial proportion of adolescents, who show an increased risk of suicide, and of developing clinical anxiety and poor mental health. Externally resourced school-based cognitive behavioural therapy (CBT) interventions have been shown to be effective in treating test anxiety. Intervening in test anxiety, a sub-clinical anxiety, may prevent anxieties from developing into a clinical disorder. The primary outcomes are test anxiety, clinical anxiety, and wellbeing, measured at baseline, post-intervention, and 6 and 12-month follow-up. In addition, to identify treatment mechanisms additional measures are taken of uncertain control, metacognition, and emotional regulation.

ELIGIBILITY:
Inclusion Criteria:

* Participants are aged 14-16 years of age
* In the upper 66th percentile of test anxiety scores

Exclusion Criteria:

* Participants are receiving other treatment for anxiety
* Participants have a diagnosis of clinical anxiety depression or Attention Deficit Hyperactivity Disorder

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Test Anxiety Inventory | Change assessed over a 12 month period
  The Test Anxiety Inventory is a 20 item measure measured on a 4-point scale (1 = Almost Never, 4 = Almost Always). Three scores are provided: Total (20 items), worry subscale (8 items) and emotionality (8 items). The total score range is 20-80 and the worry and emotionality subscale scores are 8-32. A higher score represents higher anxiety. This will administered 4 times over a 12 month period to assess change: Baseline, 6 weeks (immediate-post intervention), 6-month follow-up and 12 month follow-up.

SECONDARY OUTCOMES:
The Metacognition Questionnaire | Change assessed over a 12 month period
  The Metacognition Questionnaire is a 30-item questionnaire that consists of six subscales: Cognitive confidence, positive beliefs, cognitive self-consciousness, uncontrollability and danger, and need to control thoughts. Each subscale comprises of 5 items and uses a 4-point scale (1 = do not agree, 4 = agree very much) and the range of scores for each subscale is 5-20. A higher score represents negative beliefs about worry. These subscales will administered 4 times over a 12 month period to assess change: Baseline, 6 weeks (immediate-post intervention), 6-month follow-up and 12 month follow-up.
Cognitive Emotion Regulation Questionnaire (short version) | Change assessed over a 12 month period
  The Cognitive Emotion Regulation Questionnaire has 18 items and consists of nine subscales: Self-blame, other-blame, rumination, catastrophizing, positive refocusing, planning, positive reappraisal, putting into perspective and acceptance. Each subscale comprises of 2 items and uses a 5-point scale (1 = almost never, 5 = almost always) and the range of scores for each subscale is 2-10. A higher score represents greater use of cognitive coping strategies. These subscales will administered 4 times over a 12 month period to assess change: Baseline, 6 weeks (immediate-post intervention), 6-month follow-up and 12 month follow-up.
Motivation and Engagement Scale (uncertain control subscale) | Change assessed over a 12 month period
  4 items measure measured on a 7-point scale (1 = strongly disagree, 7 = strongly agree) resulting in a score from 7-28. A higher score represents greater uncertain control. This subscale will administered 4 times over a 12 month period to assess change: Baseline, 6 weeks (immediate-post intervention), 6-month follow-up and 12 month follow-up.
Revised Children's Anxiety and Depression Scale (panic, generalized anxiety, and social anxiety subscales) | Change assessed over a 12 month period
  The generalised anxiety subscale (6 items), panic subscale (9 items), and social anxiety subscale (9 items) of the Revised Children's Anxiety and Depression Scale, are all measured on a 4-point scale (0 = Never, 3 = Always). The range of scores for the generalised anxiety subscale is 0-18, the panic subscale is 0-27, and the social anxiety subscale is 0-27. A higher score represents higher anxiety. These subscales will administered 4 times over a 12 month period to assess change: Baseline, 6 weeks (immediate-post intervention), 6-month follow-up and 12 month follow-up.
School-related Wellbeing Scale | Change assessed over a 12 month period
  6 items measured on a 5-point scale (1 = Strongly Disagree, 5 = Strongly Agree) resulting in a score from 6-30. A higher score represents higher school-related wellbeing. These subscales will administered 4 times over a 12 month period to assess change: Baseline, 6 weeks (immediate-post intervention), 6-month follow-up and 12 month follow-up.

IPD SHARING:
Plan to Share IPD: Yes
A curated dataset will be uploaded to the Mendeley Open Data repository and assigned a doi that can be linked to all published articles via Science Direct
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be uploaded in December 2022 and remain available permanently
Access Criteria: Registration with Mendeley Open Data or Science Direct